CLINICAL TRIAL: NCT02244697
Title: The Yield of Laryngeal Ultrasound in the Evaluation of Stridor and Dysphonia in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-14-FS-0191-CTIL
Record Dates: First submitted 2014-09-02; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Stridor; Vocal Cord Paralysis
Keywords: Stridor; Vocal Cord Paralysis (VCP); Ultrasound (US)
MeSH Terms: conditions — Respiratory Sounds; Vocal Cord Paralysis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Experimental: laryngeal ultrasound stridor: Children aged 0-16 years referred for an awake nasolaryngoscopy for stridor or dysphonia at the pediatric Otolaryngology unit at the Tel Aviv Sourasky Medical Centre.
- Other: laryngeal ultrasound -control: Infants matched for age referred for ANL for reasons other than stridor will undergo US of the larynx.

SUMMARY:
Stridor is a respiratory noise caused by partial obstruction of the large airways at the level of the pharynx, larynx and/or trachea. The second most common cause of stridor is vocal cord paralysis.

Awake nasolaryngoscopyn (ANL) is regarded as the gold standard for the diagnosis of laryngomalacia. However, ANL has some drawbacks as it may cause discomfort for the patient and the laryngeal view may be obscured due to patient movement or anatomical variations.

Ultrasound (US) is a noninvasive, painless, radiation free, well tolerated imaging technique. Evaluation of the dynamic characteristics of the glottis by US revealed perfect reliability in comparison to nasolryngoscopy suggesting that US can be useful in the assessment of laryngeal adduction.

The investigator hypothesize that laryngeal US can be an accurate and reliable adjunct in the diagnosis of functional and anatomical causes of stridor and dysphonia in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

children aged 0-16 years referred for an awake nasolaryngoscopy for stridor or dysphonia at the pediatric Otolaryngology unit at the Tel Aviv Sourasky Medical Centre will undergo US of the larynx.

Exclusion Criteria:

* None

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children aged 0-16 years referred for an awake nasolaryngoscopy for stridor or dysphonia at the pediatric Otolaryngology unit at the Tel Aviv Sourasky Medical Centre will undergo US of the larynx.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
The number of participants that will be diagnosed with anatomical and functional causes of stridor and dysphonia by US in comparisom with ANL | 2014-2016
  i.e. vocal cord nodules, vocal cord paralysis, vocal cord cyst etc.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Friedman, Doctor, Principal Investigator
Locations (1):
- Sourasky Medical Centre, Tel Aviv, Israel